CLINICAL TRIAL: NCT06266429
Title: Metabolomic Profiling of Racial Disparity in Pediatric Post-tonsillectomy Pain
Brief Title: Metabolomic Profiling of Racial Disparity
Status: Active, not recruiting | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chief, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Other Study IDs: STUDY00001304
Record Dates: First submitted 2021-02-24; First posted 2024-02-20 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Adenoid Hypertrophy; Tonsillar Hypertrophy; Surgery
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood collection — Collecting blood pre-op and post-op for metabolite levels.

SUMMARY:
Tonsillectomy ± adenoidectomy (T&A) is one of the most common surgical operations with over 500,000 pediatric T&As performed annually in the United States. Unfortunately, despite advances in anesthetic and surgical techniques, moderate-severe post-tonsillectomy pain (PTP) remains a significant problem affecting up to 62% of children. PTP is thought to arise from pharyngeal mucosal inflammation, which produces local nerve irritation and pharyngeal muscle spasm. Patient factors and surgical techniques also play major roles. Race is an important phenotypic risk factor for moderately severe early PTP. The underlying molecular basis of this differential pain experience is presently unknown. This gap in knowledge means that therapies are poorly targeted and often unsuccessful. Indeed, treatment options for PTP have not advanced substantively for many years. Metabolomics provides novel opportunities to investigate common and unique "metabolic signature" of PTP through the analysis of low molecular weight compounds produced in response to tissue injury. Therefore, the central themes of this proposal are that (1) PTP is a complex process that may be determined by molecular level factors such as preoperative systemic inflammation and metabolic profile, and (2) these molecular level factors may explain the excess burden of PTP among minority children. Here the investigators seek to utilize a combined clinical, biological and untargeted metabolomics approach to identify candidate small and large serum molecules that may influence the frequency and severity of PTP in children across racial groups. This approach to exploring the molecular basis of PTP is novel and knowledge from the study should substantially enhance understanding of the mechanisms underlying pediatric PTP - and narrow the racial disparities in post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Consenting (or assenting) patients age 4-17yr and American Society of Anesthesiologist's (ASA) physical status I-III who are scheduled for elective tonsillectomy ± adenoidectomy (T&A).

Exclusion Criteria:

* Age > 18 years old
* Children below 4 years of age because they are routinely admitted following T&A in our institution and may not be able to clearly self-report their pain
* Children on chronic preoperative analgesic medications
* Children with Cushing's syndrome, or nephrotic syndrome
* Children on chronic systemic steroids
* Children with concurrent surgical procedures that could prolong the duration of anesthesia and surgery
* Children that do not speak English or cannot self-report their pain after surgery (significant cognitive impairment, anticipated or unplanned postoperative endotracheal intubation, and sedation)

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing tonsillectomy ± adenoidectomy at Nationwide Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean fold-change of metabolomics markers by race using untargeted reverse-phase liquid-chromatographic mass spectrometry | Immediately prior to surgery start and immediately post-op
  The global evaluation of small molecule biomarkers, metabolites, and the relative levels of molecular and chemical markers of post-tonsillectomy pain severity. Mass spectrometry detection following separation of protein-precipitated plasma by a C18 column liquid chromatography will provide the relative abundances of small molecule lipids, drug metabolites, amino acids, sugars, and other small potential biomarkers in subjects and using quality-control pooled analysis all samples will be normalized so that each individual metabolite can be compared between high and low-pain samples. Those metabolites found to have significant fold changes between high and low-pain subjects can be further quantified with targeted metabolomics to get absolute quantitation in plasma.
Highest pain score | Immediately after waking up from surgery
  Highest recorded post-anesthesia care unit (PACU) pain score upon emerging from general anesthesia will be assessed with the Wong-Baker face scale. Scale is 0-10, with 0 being no pain and 10 being worst pain.
Last pain score | Immediately prior to discharge
  Last recorded pain score prior to discharge from the hospital will be assessed with the Wong-Baker face scale. Scale is 0-10, with 0 being no pain and 10 being worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States